CLINICAL TRIAL: NCT04846842
Title: A Phase II Study of Gimatecan in the Treatment of Platinum-resistant Recurrent Epithelial Ovarian, Fallopian Tube or Peritoneal Cancer
Brief Title: A Study of Oral Gimatecan in Platinum-Resistant Epithelial Ovarian, Fallopian Tube or Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST1481-LEES-2020-13
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: epithelial ovarian, fallopian tube or peritoneal cancer; Platinum resistant; chemotherapy; gimatecan
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — ST 1481

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gimatecan group (Experimental): In Phase II study, patients will receive gimatecan at fixed dose level (0.8mg/m2/d, oral, every 4 weeks) until progressive disease (PD)、complete remission（CR）).
  Interventions: Drug: Gimatecan

INTERVENTIONS:
Drug: Gimatecan — Patients will receive gimatecan orally at the fixed dose level on day 1-5 every 4 weeks.
  Other Names: ST1481

SUMMARY:
This phase II clinical trial studies the safety and effect of Gimatecan in patients with platinum-resistant recurrent epithelial ovarian, fallopian tube or peritoneal cancer.

The chemotherapy will be given every four weeks.This study is a single-arm, multi-center research design.

DETAILED DESCRIPTION:
The study had 3 phases: screening phase, treatment phase and follow-up phase. During the treatment phase, the drug will continue to be administered until the progression of disease, complete remission , unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects were able to understand the informed consent, voluntarily participate in and sign the informed consent, with good compliance and cooperation with follow-up.
2. A histopathological or cytological diagnosis of epithelial ovarian, fallopian tube or peritoneal cancer.
3. Previous systematic treatment ≤ 2 lines, and progression in platinum based regimens or recurrence within 6 months after the end of platinum regimen. 1) Imaging progression of recurrence and progression should be clearly recorded;2) Neoadjuvant + adjuvant chemotherapy with platinum regimen ≥ 6 cycles, and platinum regimen after recurrence / progression ≥ 4 cycles;3) If there is progression during the treatment of platinum based regimen, the treatment cycle is not limited;4) Recurrence / progression within 6 months after the end of neoadjuvant / adjuvant therapy is considered to have received the first-line systematic treatment.
4. Measurable cancer lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
5. ≥18 years old;
6. Eastern Cooperative Oncology Group(ECOG) performance status score 0-1;
7. Estimated life expectancy >3 months;
8. The function of important organs meets the following requirements:

   1. white blood cell count (WBC) ≥ 3.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L, platelets ≥ 100×109/L, hemoglobin ≥ 90g/L;
   2. ALT, AST≤ 2.5×ULN; liver metastasis: ALT、AST≤ 5.0×ULN;
   3. serum albumin ≥ 28g/L;
   4. total bilirubin ≤ 1.5×ULN;
   5. serum creatinine ≤ 1.5×ULN, creatinine clearance rate ≥60 mL/min;
   6. PT≤ 1.5×ULN;
9. The subjects had no history of allergy to camptothecin or its components;
10. Non surgical sterilization or female subjects of childbearing age need to use a medically approved contraceptive method after signing the informed consent, during the study treatment period and within 6 months after the end of the study treatment period; non surgical sterilization female subjects of childbearing age must have negative blood HCG test within 3 days before entering the study; and they must be in non lactation period.
11. Taking drugs orally;
12. The subjects had recovered and treatment will start more than 4 weeks after the end of previous surgery, chemotherapy, targeted therapy and radiotherapy.

Exclusion Criteria:

1. Subjects who have been treated previously with topotecan, Irinotecan or other topoisomerase I inhibitors;
2. Other anticancer therapy including any investigational agent within 30 days prior to the first dose of the investigational drug gimatecan;
3. Within 14 days before the first dose of the investigational drug gimatecan, any active infection requiring systemic anti infective treatment;
4. Subjects with a history of major gastrointestinal surgery (e.g., total gastrectomy, small bowel resection) or gastrointestinal dysfunction that may alter drug absorption and activity in vivo;
5. Severe cardiovascular disease, such as NYHA grade 3-4 heart failure;
6. Patients who have been treated previously with intravenous or oral drugs that affect CYP isoenzymes within 7 days prior to the first dose of the investigational drug gimatecan;
7. A history of immunodeficiency (including a positive HIV test result);Presence of active hepatitis B , hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay);
8. Pleural effusion, pericardial effusion or ascites with clinical symptoms can not be controlled by puncture drainage or other treatment;
9. Subjects with hereditary or acquired bleeding tendency (hemophilia, thrombocytopenia, etc.), interstitial pneumonia or pulmonary fibrosis, and active tuberculosis (whether or not treated) in the past year;
10. Vaccinated with live attenuated vaccine within 4 weeks;
11. Subjects had other active malignancies within 5 years before the first dose of the investigational drug gimatecan;
12. Subjects with active meningeal metastasis or uncontrollable and untreated brain metastasis.
13. Other considered unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | To evaluate objective response rate every 8 weeks after the initiation of chemotherapy, up to 24 months.
  Percentage of patients with objective response assessed by best overall response (BOR) and independent review committee （IRC） of either complete response(CR) or partial remission(PR) will be reported.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year progression free survival of the whole group.
Disease control rate (DCR) | To evaluate disease control rate every 8 weeks after the initiation of chemotherapy, up to 24 months.
  will be reported.
Duration of Response (DoR) | From date of randomization until the date of death from any cause or the date of last follow-up whichever came first, assessed up to 24 months.
  The 2-year overall survival of the whole group.
Overall survival (OS) | From date of randomization until the date of death from any cause or the date of last follow-up whichever came first, assessed up to 24 months.
  The 2-year overall survival of the whole group.

CONTACTS AND LOCATIONS:
Overall Officials: ZHOU QI, Study Director — Chongqing Tumor Hospital

REFERENCES:
- [Result] Hurwitz JL, McCoy F, Scullin P, Fennell DA. New advances in the second-line treatment of small cell lung cancer. Oncologist. 2009 Oct;14(10):986-94. doi: 10.1634/theoncologist.2009-0026. Epub 2009 Oct 9. PMID 19819917